CLINICAL TRIAL: NCT03058822
Title: A Randomized, Open-label, Parallel-group, Single Subcutaneous Dose, Relative Bioavailability Study of the Pharmacokinetics of Lulizumab (BMS-931699) From Prefilled Syringe (Process A) Compared to Drug in Vial (Process A) in Healthy Participants
Brief Title: Relative Bioavailability of BMS-931699 From Prefilled Syringe Compared to Drug in Vial
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business objectives have changed
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IM128-037
Record Dates: First submitted 2017-01-10; First posted 2017-02-23 (Actual); Last update posted 2017-12-20 (Actual); Status verified 2017-12

CONDITIONS: Healthy
MeSH Terms: interventions — lulizumab pegol

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Prefilled Syringe Upper Arm (Experimental): Single subcutaneous dose from prefilled syringe into upper arm of BMS-931699
  Interventions: Drug: BMS-931699
- Prefilled Syringe Thigh (Experimental): Single subcutaneous dose from prefilled syringe into thigh of BMS-931699
  Interventions: Drug: BMS-931699
- Prefilled Syringe Abdomen (Experimental): Single subcutaneous dose from prefilled syringe into abdomen of BMS-931699
  Interventions: Drug: BMS-931699
- Drug in Vial Upper Arm (Experimental): Single subcutaneous dose from drug in vial into upper arm of BMS-931699
  Interventions: Drug: BMS-931699
- Drug in Vial Thigh (Experimental): Single subcutaneous dose from drug in vial into thigh of BMS-931699
  Interventions: Drug: BMS-931699
- Drug in Vial Abdomen (Experimental): Single subcutaneous dose from drug in vial into abdomen of BMS-931699
  Interventions: Drug: BMS-931699

INTERVENTIONS:
Drug: BMS-931699 — BMS-931699 single subcutaneous dose on Day 1

SUMMARY:
A Phase 1, relative bioavailability study of BMS-931699 from prefilled syringe compared to drug in vial

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants as determined by no clinically significant deviation from normal in medical history, physical examination, electrocardiograms, and clinical laboratory determinations
* All participants must have hemoglobin, hematocrit, and platelets within normal limits at screening
* All participants must have activated partial thromboplastin time, prothrombin time, and international normalized ratio within normal limits at screening

Exclusion Criteria:

* Any current or past history or risk for tuberculosis:
* Active tuberculosis requiring treatment within the previous 3 years. All participants will be required to have a QuantiFERON tuberculosis Gold or T-SPOT tuberculosis test performed at screening. Also excluded are participants with evidence of a past tuberculosis infection without documented adequate therapy. Participants with a positive QuantiFERON tuberculosis Gold or T-SPOT tuberculosis test at screening will not be eligible for the study. A QuantiFERON tuberculosis Gold or T-SPOT tuberculosis test performed within 4 weeks of dosing on Day 1 is acceptable as long as there is documentation of a negative result.
* Current clinical, radiographic, or laboratory evidence of active tuberculosis
* A history of herpes zoster

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2017-01-25 (Actual); Primary Completion 2017-03-30 (Actual); Study Completion 2017-03-30 (Actual)

PRIMARY OUTCOMES:
Relative bioavailability of BMS-931699 following a single subcutaneous dose from prefilled syringe relative to drug in vial in healthy participants | 43 days

SECONDARY OUTCOMES:
Safety and tolerability of BMS-931699 following a single prefilled syringe or drug in vial subcutaneous dose in healthy participants by assessing adverse events and other physical assessments throughout study conduct | 43 days

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Qps-Mra, Llc, South Miami, Florida, United States

REFERENCES:
- See also: BMS Clinical Trial Education Resource — http://www.bms.com/studyconnect/pages/home.aspx
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/pages/investigator_inquiry_form.aspx
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/Recalls/